CLINICAL TRIAL: NCT06422130
Title: Ningbo Maternity-Child Linked Database Study(MATCHLESS): Using Electronic Health Records to Improve Maternal and Child Health Care and Outcomes in China
Brief Title: Ningbo Maternity-Child Linked Database Study
Acronym: MATCHLESS
Status: Active, not recruiting | Type: Observational
Sponsor: Ningbo University (Other)
Collaborators: Ningbo Health Information Center (Unknown)
Responsible Party: Principal Investigator, Liya Liu, Associate Professor, Ningbo University
Other Study IDs: NBU-2023-240
Record Dates: First submitted 2024-05-08; First posted 2024-05-20 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Pregnant Women; Children
Keywords: Population-based healthcare database; Longitudinal study; Ambispective Cohort; Pregnant women and offspring
MeSH Terms: interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women and their offspring
  Interventions: Other: Pregnant women and their offspring without intervention

INTERVENTIONS:
Other: Pregnant women and their offspring without intervention — Pregnant women and their offspring with those exposures of interest determined in specific research based on the database

SUMMARY:
With the implementation of China's two-child policy and a marked increase in adverse pregnancy outcomes, leveraging electronic health records (EHR) to enhance maternal and child healthcare and outcomes in China has emerged as a novel strategy to tackle this pivotal demographic and health challenge. Given the mature construction of the information platform and the well-established maternal and child health service system in Ningbo, this study utilized the Ningbo Maternal and Child Health Electronic Monitoring Information Management System and the Ningbo Regional Health Information Platform to conduct the Ningbo maternity-child linked database study (MATCHLESS), which involved over 300,000 mother-child pairs in China. MATCHLESS not only allows for longitudinal follow-up of pregnant women and their offspring but also expands its scope from prenatal exposure to long-term outcomes through data linkage. The longitudinal scope of MATCHLESS facilitates the elucidation of the relationship and etiological significance of early-life exposures and adverse pregnancy outcomes. It also permits the exploration of the health trajectory of women and children over their life-course.

During the past 5 years (October 2016 to December 2021), a substantial amount of maternal and child health data has been recorded in MATCHLESS, including socio-demographics, health care services and medications, as well as clinical outcome events. Additionally, it contains longitudinal measurements on risk factors for adverse pregnancy outcomes, which provides a robust foundation for future real-world studies of dynamic predictive models. This study was approved by the Ethics Review Committee of the Ningbo University Health Science Center. Considering the safety, privacy, and confidentiality concerns surrounding the storage and processing of personal EHR data, the responsibility for data storage and management is undertaken by the Health Commission of Ningbo. Researchers are required to submit applications to the local health department, and all studies undergo ethical review and research registration procedures to access EHR data for health research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women and their offspring who registered at the Ningbo maternal and child health electronic monitoring information management system.

Exclusion Criteria:

* None.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — All pregnant women and their offspring registered at the Ningbo maternal and child health electronic monitoring information management system were enrolled.
Study Population: Pregnant women and their offspring who registered at the Ningbo maternal and child health electronic monitoring information management system.
Sampling Method: Non-Probability Sample
Enrollment: 325596 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of preterm birth | Up to 42 weeks
  Regular contractions accompanied by cervical change at less than 37 weeks' gestation.
  Or, the following diagnose in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : O60.
Incidence of pre-eclampsia | Up to 42 weeks
  New onset hypertension (>140 mm Hg systolic or >90 mm Hg diastolic) after 20 weeks of pregnancy and the coexistence of one or both of the following new-onset conditions: proteinuria (urine protein:creatinine ratio ≥30 mg/mmol, or albumin: creatinine ratio ≥8 mg/mmol, or ≥1 g/L [2+] on dipstick testing), other maternal organ dysfunction, including features such as renal or liver involvement, neurological or haematological complications, or uteroplacental dysfunction (such as fetal growth restriction, abnormal umbilical artery Doppler waveform analysis, or stillbirth).
  Or, the following diagnose in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : O14.
Incidence of eclampsia | Up to 42 weeks
  The occurrence of new-onset, generalized, tonic-clonic seizures or coma in a patient with preeclampsia or gestational hypertension.
  Or, the following diagnose in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : O15.
Incidence of gestational diabetes mellitus | Up to 42 weeks
  Impaired Glucose Tolerance (IGT) with onset or first recognition during pregnancy.
  Or, the following diagnose in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : O24.4.
Incidence of low birth weight | Up to 42 weeks
  Weight at birth of < 2500 g.
  Or, at least one of the following diagnoses in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : P07.0, P07.1.
Incidence of small for gestational age | Up to 42 weeks
  Less than the tenth birth weight centile using INTERGROWTH-21st.
  Or, the following diagnose in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : P05.
Incidence of autism | Up to 10 years
  The following diagnose in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : F84.
Incidence of birth defects | Up to 10 years
  Birth defects such as congenital malformations of the nervous system, congenital malformations of eye, ear, face and neck, congenital malformations of the circulatory system, congenital malformations of the respiratory system, or other birth defects.
  Or, at least one of the following diagnoses in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : Q00-Q99.
Incidence of postpartum hemorrhage | Within 24 hours after delivery
  Blood loss exceeding 500 mL following vaginal birth and 1000 mL following cesarean.
  Or, the following diagnose in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : O72.
Incidence of stillbirth | Up to 42 weeks
  Death of a fetus that has reached a birth weight of 500 g, or if birth weight is unavailable, gestational age of 22 weeks or crown-to-heel length of 25 cm.
  Or, at least one of the following diagnoses in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : Z37.1, Z37.3, Z37.4, Z37.7.
Incidence of ruptured uterus | Up to 42 weeks
  Uterine rupture is confirmed by laparotomy.
  Or, at least one of the following diagnoses in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : O71.0, O71.1, O34.5, O62.4.
Incidence of maternal death | Up to 52 weeks
  Death of women while pregnant or within 42 days of termination of pregnancy irrespective of the site and size of pregnancy but related to or aggravated by the pregnancy or its management but not from accidental or incidental causes.
Incidence of neonatal death | Within 28 days after delivery
  Deaths among live births during the first 28 completed days of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo University, Ningbo, Zhejiang, China

REFERENCES:
- [Derived] Li N, Ye H, Zhu H, Liang M, Wang K, Zhao Y, Liu L. Association of prenatal exposure to air pollution with autism spectrum disorder: A population-based retrospective cohort study in China. Environ Res. 2026 Feb 15;291:123612. doi: 10.1016/j.envres.2025.123612. Epub 2025 Dec 22. PMID 41443491